CLINICAL TRIAL: NCT00497159
Title: A Multi-Center, Phase 2 Randomized, Double-Blinded, Placebo-Controlled Study of Dimebon in Subjects With Huntington's Disease
Brief Title: A Study of the Novel Drug Dimebon in Patients With Huntington's Disease
Acronym: DIMOND
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medivation, Inc. (Industry)
Collaborators: Huntington Study Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DIM05
Record Dates: First submitted 2007-07-03; First posted 2007-07-06 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-05

CONDITIONS: Huntington's Disease
Keywords: Trial of Dimebon to treat patients with mild-to-moderate Huntington's disease.
MeSH Terms: conditions — Huntington Disease | interventions — latrepirdine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator): Placebo
  Interventions: Other: Placebo
- 2 (Experimental): Dimebon
  Interventions: Drug: Dimebon

INTERVENTIONS:
Other: Placebo — Placebo TID x 90 days
  Arms: 1
Drug: Dimebon — Dimebon 20 mg TID x 90 days
  Arms: 2

SUMMARY:
This study will evaluate the safety of 3 months of Dimebon dosing and the efficacy of Dimebon in improving cognitive, motor, and overall function in subjects with Huntington's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Clinical features of HD and a confirmatory family history of HD, and/or genetically confirmed HD;
* Able to take medication (capsules) by mouth.

Exclusion Criteria:

* Clinical evidence of unstable medical illness;
* Females who are pregnant or lactating or who intend to become pregnant during the study period.

Min Age: 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2007-07; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of Dimebon during 3 months of treatment in subjects with Huntington's Disease. | 90 days

SECONDARY OUTCOMES:
To assess the impact of Dimebon during 3 months of treatment on cognitive, motor, and overall function in subjects with Huntington's Disease. | 90 days
To assess the pharmacokinetics of Dimebon. | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Karl Kieburtz, MD, MPH, Principal Investigator — Huntington Study Group, University of Rochester
Locations (1):
- Huntington Study Group, Rochester, New York, United States

REFERENCES:
- [Derived] Kieburtz K, McDermott MP, Voss TS, Corey-Bloom J, Deuel LM, Dorsey ER, Factor S, Geschwind MD, Hodgeman K, Kayson E, Noonberg S, Pourfar M, Rabinowitz K, Ravina B, Sanchez-Ramos J, Seely L, Walker F, Feigin A; Huntington Disease Study Group DIMOND Investigators. A randomized, placebo-controlled trial of latrepirdine in Huntington disease. Arch Neurol. 2010 Feb;67(2):154-60. doi: 10.1001/archneurol.2009.334. PMID 20142523
- See also: The Huntington Study Group is a non-profit group of physicians and health care providers from medical centers in the US, Canada, Europe, and Australia, experienced in the care of HD patients and dedicated to clinical research of HD. Click for more info. — http://www.huntington-study-group.org